CLINICAL TRIAL: NCT00944931
Title: High-Density Direct Current Brain Polarization
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 090196; 09-N-0196
Record Dates: First submitted 2009-07-22; First posted 2009-07-23 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2012-02-09

CONDITIONS: Healthy Volunteer; HV
Keywords: Cerebral Cortex; Cognition; Motor Cortex; Cognitive Enhancement; Prefrontal Cortex; Healthy Volunteer

INTERVENTIONS:
Device: DC Brain Polarization

SUMMARY:
Background:

* Direct current (DC) brain polarization is a technique in which very weak electricity is applied to the head. Doctors have used DC polarization for many years on patients and healthy people with no known serious side effects. Earlier, researchers found that DC polarization can temporarily improve the ability of healthy people to think of certain words.
* A disadvantage of existing methods of DC polarization is that they use large electrodes and the current spreads over a large area of the brain. This makes it difficult to target particular brain areas. High-density DC polarization uses several small electrodes to focus the current in a small area of the brain. This study will test high-density DC polarization for the first time in humans.

Objectives:

* To see how well high-density direct current polarization works in the brain.
* To test a new method of performing direct current brain polarization.

Eligibility:

- Healthy, right-handed adults, ages 18 and older, who have no history of neurological or psychiatric illnesses.

Design:

* After an initial screening visit with clinical examination, participants may be assigned to one or both experiments of the study.
* Experiment 1: Participants will have electrodes placed on the left side of their heads, and will be asked to say aloud as many words as they can think of that begin with certain letters. After the high-density DC polarization current is turned on and run for 10 minutes, participants will say words beginning with a different set of letters and perform reaction time and thinking speed tests. Some participants will receive real polarization and others will not, although all participants will be told that they are receiving the polarization.
* Experiment 2: Participants will have DC brain polarization performed with transcranial magnetic stimulation (TMS), which uses magnetic pulses to activate nerve cells in the brain. We will use TMS to help us understand how far the effect of DC polarization spreads in the brain. After attaching electrodes to a point on the scalp above the ear, researchers will give about 50 TMS pulses to five different places near this area. These pulses will produce some painless muscle twitches in the hand or arm. The TMS pulses will be followed by the DC brain polarization, and then by another set of TMS pulses to see if there are any differences in muscle response.

DETAILED DESCRIPTION:
Objective:

The principal objectives are: 1) to explore the effectiveness of anodal high-density direct current (HDDC) stimulation of the brain; and 2) test the focality of the technique.

Study Population:

Up to 81 healthy volunteers over the age of 18 will be enrolled.

Design:

We will perform three studies:

1. A parallel trial of anodal and sham HDDC delivered to the lateral prefrontal area,
2. An exploratory evaluation of the focality of HDDC in the motor cortex and
3. A study to determine whether HDDC can be better targeted using a finite element model (FEM) based on the individual subject's MRI scan (obtained as part of the study).

Outcome Measures:

The primary outcome measures are the effect of anodal HDDC (relative to sham) on category verbal fluency, and the decay in the HDDC-induced change in corticospinal output excitability with distance from the active electrode. Performance on the California Computerized Assessment Package is included as a secondary safety outcome.

ELIGIBILITY:
* INCLUSION CRITERIA:

Healthy volunteers over age 18

EXCLUSION CRITERIA:

Any history of central nervous system illness or behavioral disorder

Broken skin or other lesions in the area of the electrodes

Uncontrolled medical problems, such as diabetes mellitus, hypertension, pulmonary or airway disease, heart failure, coronary artery disease, or any other condition that poses a risk for the subject during participation or potentially worsen the outcome of a burn

Presence of metal in the cranial cavity

Holes in the skull made by trauma or surgery

Pacemakers, medication pumps, and other implanted electronic hardware

Pregnancy (female volunteers who have the potential to become pregnant will have urine pregnancy test performed within 24 hours of participation)

Left handers will be excluded from Experiment 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-07-20; Primary Completion 2011-04-05 (Actual); Study Completion 2011-04-05 (Actual)

PRIMARY OUTCOMES:
Verbal fluency; focality of effect on MEP (exploratory)

CONTACTS AND LOCATIONS:
Overall Officials: William H Theodore, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Bikson M, Radman T, Datta A. Rational modulation of neuronal processing with applied electric fields. Conf Proc IEEE Eng Med Biol Soc. 2006;2006:1616-9. doi: 10.1109/IEMBS.2006.259548. PMID 17946911
- [Background] BINDMAN LJ, LIPPOLD OC, REDFEARN JW. Long-lasting changes in the level of the electrical activity of the cerebral cortex produced bypolarizing currents. Nature. 1962 Nov 10;196:584-5. doi: 10.1038/196584a0. No abstract available. PMID 13968314
- [Background] CREUTZFELDT OD, FROMM GH, KAPP H. Influence of transcortical d-c currents on cortical neuronal activity. Exp Neurol. 1962 Jun;5:436-52. doi: 10.1016/0014-4886(62)90056-0. No abstract available. PMID 13882165